CLINICAL TRIAL: NCT01228396
Title: A Randomised, Double-blind, Placebo-controlled Study of AIMSPRO in Treating Bladder Dysfunction in Secondary Progressive Multiple Sclerosis
Brief Title: AIMSPRO in the Treatment of Bladder Dysfunction in Secondary Progressive Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daval International Limited (Industry)
Responsible Party: Dr. Bryan Youl, Daval International Limited
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIMS04
Record Dates: First submitted 2010-09-26; First posted 2010-10-26 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: bladder; optic neuritis; secondary progressive multiple sclerosis; AIMSPRO; hyperimmune caprine serum; hyperimmune goat serum
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Optic Neuritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hyperimmune caprine serum against HIV lysate — 1.0ml solution for subcutaneous injection (4.5mg total protein / ml) twice weekly for 4 weeks
  Other Names: AIMSPRO

SUMMARY:
Patients with marked bladder dysfunction as a result of secondary progressive multiple sclerosis are being recruited to receive AIMSPRO or placebo by subcutaneous injection, in this double-blind crossover study.

DETAILED DESCRIPTION:
Treatment periods of 4 weeks' duration are separated by a 6 week wash-out phase. After 14 weeks of randomised therapy there is a 38 week period of "open-label" AIMSPRO treatment.

ELIGIBILITY:
Inclusion Criteria:

* M / F aged 18 years or older.
* Patients of childbearing potential must use adequate birth control measures for the duration of the study and 6 months after receiving the last injection of AIMSPRO.
* Clinically definite SPMS.
* Ambulant, walking aids allowed.
* No more than one relapse within the last 12 months and no relapse within the last 6 months.
* Urinary frequency of at least 8 times per 24-hours.
* Urinary urgency with or without urge incontinence.
* MRI brain or spinal cord abnormalities consistent with MS.
* Screening laboratory test results must meet the following criteria:

  * Haemoglobin > 9.5 g/dL
  * WBC > 3.5 x 109/L
  * Neutrophils > 1.5 x 109/L
  * Platelets > 100 x 109/L
* Baseline AST , alkaline phosphatase, Thyroid function, Serum Electrophoresis levels must be within the normal range.
* Able to adhere to the study visit schedule and other protocol requirements
* Capable of giving written informed consent.

Exclusion Criteria:

* Acute symptomatic urinary infection.
* Taking DDAVP or antimuscarinic agents.
* Full time wheelchair user.
* Immunosuppressant drug therapy of any kind in the last 3 months.
* Relapse within the last 6 months.
* No clear progression of disability in the last 12 months.
* Co-existent medical condition precluding participation, including any history of severe allergic reaction.
* Pregnant or lactating women and women who are planning pregnancy within 12 months of screening (i.e., approximately 6 months following last injection).
* Receipt of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Treatment with any therapeutic agent targeted at reducing TNF (e.g., infliximab, pentoxifylline, thalidomide, etanercept, etc.) within 3 months of screening.
* Previous administration of AIMSPRO.
* Ongoing corticosteroid therapy or any corticosteroids within the previous 3 months.
* History of known allergy to animal proteins, tuberculosis.
* Serious infections (such as pneumonia or pyelonephritis) in the previous 3 months. Less serious infections such as acute upper respiratory tract infection or simple urinary tract infection, should be followed to their conclusion or treated, as appropriate, prior to inclusion.
* Patients with opportunistic infections within the previous 6 months.
* Established malignant disease, renal, hepatic, haematologic, gastrointestinal, endocrine, pulmonary, or cardiac disease.
* Significant other neurological disorder.
* Presence of a transplanted organ, with the exception of a corneal transplant > 3 months prior to screening.
* Lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Recent clinically significant substance abuse (drug or alcohol).
* Poor tolerability of venipuncture.
* Investigational drugs or drugs targeted at reducing TNF are not allowed during participation in the study.
* Patients will not be permitted to receive immunosuppressive treatment during this study. The exception will be where a patient's treating neurologist determines that a course of steroid therapy, oral or intravenous, is required in view of a sufficiently disabling relapse of MS.
* Immunosuppressive therapy within the month prior to entry into the study.
* Taking the licensed anticonvulsant medication lamotrigine or the anti-arrhythmic drug flecainide, both of which are potent sodium channel blocking agents.
* Unable to fill in the criteria related to bladder dysfunction status.
* Unable to give written informed consent.
* Use of intermittent or indwelling urinary catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in average voided volume | At 0, 4, 10 and 14 weeks
  The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.

SECONDARY OUTCOMES:
Change in average 24-hour frequency | At 0, 4, 10 and 14 weeks
  The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in visual acuity and colour vision | At 0, 4, 10 and 14 weeks
  Employs logMAR based and Farnsworth-Munsell 100 Hue testing. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in average 24-hour incontinence | At 0, 4, 10 and 14 weeks
  The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in urgency score | At 0, 4, 10 and 14 weeks
  The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in I-QOL score | At 0, 4, 10 and 14 weeks
  The Incontinence - Quality of Life questionnaire is administered at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in Whittington Urgency Score | At 0, 4, 10 and 14 weeks
  The Whittington Urgency Score is administered at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in Kurtzke EDS | At 0, 4, 10 and 14 weeks
  The Kurtzke EDS assessment is undertaken at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in MSIS-29 | At 0, 4, 10 and 14 weeks
  The Multiple Sclerosis Impact Scale is administered at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in MS FC | At 0, 4, 10 and 14 weeks
  The The Multiple Sclerosis Functional Composite assessment is undertaken at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.
Change in MS WS | At 0, 4, 10 and 14 weeks
  The Multiple Sclerosis Walking Scale is assessed at the beginning and end of each four week treatment phase. The change is calculated as the value at the later time point minus the value at the earlier time point for weeks 0 to 4 and weeks 10 to 14 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: James Malone-Lee, MD, Principal Investigator — University College, London
Locations (1):
- Royal Free Hospital Hampstead NHS Trust, London, United Kingdom